CLINICAL TRIAL: NCT04888312
Title: An Open-label Phase 1b/2 Study Assessing the Safety and Efficacy of Mitazalimab in Combination With Chemotherapy in Patients With Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Safety and Efficacy of Mitazalimab in Combination With Chemotherapy in Pancreatic Cancer Patients
Acronym: OPTIMIZE-1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alligator Bioscience AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-20-1013-C-03
Record Dates: First submitted 2021-05-06; First posted 2021-05-17 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: mitazalimab; modified FOLFIRINOX; Pancreatic ductal adenocarcinoma; PDAC; Pancreatic Cancer; Chemotherapy, combination; 5-Fluorouracil; Oxaliplatin; Leucovorin; Irinotecan
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy; mitazalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intravenously administered mitazalimab given in combination with chemotherapy (Experimental): Mitazalimab, a human monoclonal antibody targeting CD40, administered intravenously every 14 days, in combination with standard of care chemotherapy modified FOLFIRINOX.
  Interventions: Biological: CD40 agonist mitazalimab in combination with chemotherapy

INTERVENTIONS:
Biological: CD40 agonist mitazalimab in combination with chemotherapy — Mitazalimab administered intravenously every 14 days in combination with standard of care chemotherapy modified FOLFIRINOX.
  Other Names: ADC-1013, JNJ-64457107

SUMMARY:
Phase 1b/2 study to assess the safety and efficacy of mitazalimab in combination with chemotherapy in patients with metastatic pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
OPTIMIZE-1 is a phase 1b/2, open-label, multi-center study assessing the clinical efficacy of mitazalimab in combination with chemotherapy in patients with metastatic pancreatic ductal adenocarcinoma.

The efficacy of intravenously administered mitazalimab in combination with the standard of care chemotherapy mFOLFIRINOX will be evaluated in patients with metastatic pancreatic ductal adenocarcinoma. Two dose levels of mitazalimab, 450 ug/kg and 900 ug/kg, are planned to be evaluated together with mFOLFIRINOX for determination of recommended phase 2 dose (RP2D) of mitazalimab in combination with mFOLFIRINOX before entering a dose expansion part with RP2D obtained. The expansion part will evaluate the clinical efficacy of mitazalimab in combination with mFOLFIRINOX assessing objective response rate (ORR), primary endpoint, as well as Progression-free survival (PFS) and Overall survival (OS). The dose expansion part includes a Simon´s two-stage design with an interim analysis for stop for futility or efficacy based on ORR.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent
2. Is ≥18 years of age at the time of signing the informed consent form (ICF)
3. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Has a diagnosis of previously untreated metastatic pancreatic ductal adenocarcinoma (histologically documented)
5. Has measurable disease per RECIST v. 1.1
6. Has not received previous chemotherapy for pancreatic ductal adenocarcinoma
7. Has not received prior abdominal radiotherapy (except for palliative radiotherapy to non-target lesions)
8. Has a life expectancy of ≥ 3 months
9. Has acceptable hematologic laboratory values defined as:

   1. Neutrophils ≥ 1.5 x 109/L without growth factor stimulation within 3 weeks prior to the blood test
   2. Platelets ≥100 x 109/L
   3. Hemoglobin ≥6.2 mmol/L (~100 g/L) (may be after transfusion)
10. Has acceptable clinical chemistry laboratory values defined as:

    1. Bilirubin ≤1.5 x ULN (biliary drainage is permitted)
    2. AST ≤3 x ULN (irrespective of hepatic metastases)
    3. ALT ≤3 x ULN (irrespective of hepatic metastases)
    4. Creatinine ≤1.5 x ULN or glomerular filtration rate (GFR) of ≥45 mL/min
    5. INR ≤1.5 x ULN
    6. Albumin ≥28 g/L
11. For women of childbearing potential1:

    1. Has a negative highly sensitive serum (β-human chorionic gonadotropin [β-hCG]) pregnancy test at screening
    2. Is willing to use highly effective contraception methods during study treatment and for at least six months thereafter
12. Fertile men must practice effective contraceptive methods (i.e. surgical sterilization, or a condom used with a spermicide) during study treatment and for at least six months thereafter
13. Is willing to comply with all study procedures

Exclusion Criteria:

1. Has other types of non-ductal tumor of the pancreas, including endocrine tumors or acinar cell adenocarcinoma, cyst adenocarcinoma and ampullary carcinoma
2. Has other current cancer or history of cancer in the prior 3 years before signing the ICF other than in situ cervical cancer, or basal cell or squamous cell carcinoma treated with local excision only
3. Has known CNS metastases or carcinomatous meningitis
4. Has contraindication to any constituent of study treatment (mitazalimab and applicable chemotherapy)
5. Has a history of chronic diarrhea, inflammatory disease of the colon or rectum, or unresolved partial or complete intestinal obstruction
6. Has a history of myocardial infarction within 12 months of the first administration of mitazalimab, uncontrolled angina pectoris, unstable cardiac arrhythmias, or congestive heart failure of New York Heart Association class II or greater
7. Has QTc >450 msec
8. Has uncontrolled intercurrent illness, including active infection
9. Has a known history of HIV, hepatitis B or active hepatitis C infection
10. Is a female patient who is pregnant or nursing
11. Has received attenuated vaccine within 28 days before the first dose of study treatment
12. Any condition that, in the opinion of the Investigator, would place the patient at increased risk or preclude the patient's compliance with the study
13. Participates in another investigational drug or device study with any intervention within the previous 4 weeks prior to first dose of mitazalimab
14. Has received prior treatment with irinotecan or platinum-containing chemotherapy
15. Has pre-existing peripheral neuropathy greater than grade 1
16. Has known Gilbert's disease
17. Has known genotype UGT1A1 * 28 / * 28
18. Has known fructose intolerance (malabsorption)
19. Has complete dihydropyrimidine dehydrogenase (DPD) deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) (Part 1: Phase 1b Dose escalation) | From first dose to end of dose limiting toxicity period (Day 1-21)
  Number of patients experiencing DLTs
Objective response rate (ORR) (Part 2: Phase 2 Dose expansion) | From first dose to 28-56 days after end of study treatment
  Proportion of patients achieving complete response or partial response at any time during the study

SECONDARY OUTCOMES:
Type, frequency and severity of Adverse Events | From informed consent signed to 28-56 days after end of of study treatment
  Number of patients experiencing AEs. Number of events summarized by SOC and preferred term.
Anti-drug-antibody (ADA) titer in serum (tolerability) | From first dose until 28-56 days after end of study treatment
  Immunogenicity of mitazalimab
Cmax of mitazalimab (pharmacokinetics) | From first dose until 28-56 days after end of study treatment
  Cmax derived from mitazalimab serum concentrations
Tmax of mitazalimab (pharmacokinetics) | From first dose until 28-56 days after end of study treatment
  Tmax derived from mitazalimab serum concentrations
AUC(0-T) of mitazalimab (pharmacokinetics) | From first dose until 28-56 days after end of study treatment
  AUC(0-T) derived from mitazalimab serum concentrations
Anti-tumor Activity per RECIST 1.1 guideline (efficacy) | From first dose until 28-56 days after end of study treatment
  Best overall response, duration of response, Duration of stable disease, disease control rate, Time to next anti-cancer therapy will be assessed
Progression free survival (efficacy) | From first dose and up to 2 years after end of study treatment
  Number of days from first dose of mitazalimab to progressive disease or death.
Overall survival (efficacy) | From first dose and up to 2 years after end of study treatment
  Number of days from first dose of mitazalimab until death

CONTACTS AND LOCATIONS:
Overall Officials: Yago Pico de Coaña, PhD, Study Director — Alligator Bioscience AB; Jean-Luc van Laethem, Prof. MD, Principal Investigator — Hospital Erasme
Locations (14):
- Belgium (4):
  - Cliniques Universitaires St-Luc, Brussels
  - Hospital Erasme, Brussels
  - UZA Antwerp, Edegem
  - Universitair Ziekenhuis Gent, Ghent
- France (5):
  - Centre Hospitalier Universitaire de Bordeaux - Hôpital Haut-Lévêque,, Bordeaux
  - Centre Lyon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Hopital Européen Georges Pompidou, Paris
  - Institute de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
- Spain (5):
  - Hospital Universitario Vall d'Hebron, Barcelona, Spain, Barcelona
  - Hospital Universitario La Paz, Madrid, Spain, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid, Spain, Madrid
  - Hospital Universitario Virgen del Rocio, Sevilla, Spain, Seville
  - Hospital Universitario Miguel Servet, Zaragoza, Spain, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Laethem JL, Geboes K, Borbath I, Macarulla Mercade T, Lambert A, Cassier P, Prenen H, Mitry E, Blanc JF, Pilla L, Feliu J, Rodriguez Garrote M, Pazo-Cid RA, Gallego I, Smith KE, Nordbladh K, Jimenez DG, Ellmark P, Pico de Coana Y, Ambarkhane SV, Beatty GL, O'Reilly EM. CD40 agonist mitazalimab with mFOLFIRINOX in untreated metastatic pancreatic cancer: Biomarkers associated with outcomes from OPTIMIZE-1. Cell Rep Med. 2025 Oct 21;6(10):102407. doi: 10.1016/j.xcrm.2025.102407. Epub 2025 Oct 7. PMID 41061701
- [Derived] Van Laethem JL, Borbath I, Prenen H, Geboes KP, Lambert A, Mitry E, Cassier PA, Blanc JF, Pilla L, Batlle JF, Garrote MR, Pazo-Cid RA, Gallego I, Smith KE, Ellmark P, Pico de Coana Y, Ambarkhane SV, Macarulla T. Combining CD40 agonist mitazalimab with mFOLFIRINOX in previously untreated metastatic pancreatic ductal adenocarcinoma (OPTIMIZE-1): a single-arm, multicentre phase 1b/2 study. Lancet Oncol. 2024 Jul;25(7):853-864. doi: 10.1016/S1470-2045(24)00263-8. Epub 2024 Jun 1. PMID 38834087